CLINICAL TRIAL: NCT05040802
Title: Effectiveness of Adacel Vaccination in Pregnancy at Preventing Pertussis in Infants < 2 Months of Age in the United States (US)
Brief Title: Effectiveness of Adacel Vaccination in Pregnancy at Preventing Pertussis in Infants < 2 Months of Age in the United States
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: TD500059
Record Dates: First submitted 2021-09-07; First posted 2021-09-10 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-04

CONDITIONS: Pertussis (Whooping Cough)
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pertussis Case Group: Infants between 2 days to less than 2 months of age for whom a case of pertussis was reported (laboratory confirmed pertussis, epidemiological linkage to a laboratory-confirmed case and/or clinically compatible illness) and who met case inclusion criteria.
  This post-hoc analysis was limited to infants born of mothers vaccinated with Adacel or who did not receive any tetanus, diphtheria, and acellular pertussis (Tdap) vaccine.
  Interventions: Other: Not applicable / dataset analysis
- Control Group: Infants born at the same hospital as the case-infant who were less than 2 months old on the case-infant's cough onset date, and who met control inclusion criteria.
  This post-hoc analysis was limited to infants born of mothers vaccinated with Adacel or who did not receive any Tdap vaccine.
  Interventions: Other: Not applicable / dataset analysis

INTERVENTIONS:
Other: Not applicable / dataset analysis — Not applicable / dataset analysis

SUMMARY:
The purpose of this study is to determine the effectiveness of Adacel against pertussis disease in infants < 2 months when administered during pregnancy following the current Advisory Committee on Immunization Practices (ACIP) recommendations, i.e., from 27 to 36 weeks of gestation, and 14 days or more before delivery.

DETAILED DESCRIPTION:
The original study included cases recorded from 01 January 2011 through 31 December 2014, based on retrospective case-control methodology.

ELIGIBILITY:
Inclusion Criteria:

Cases were included if they met the following inclusion criteria:

* Reported pertussis disease in the referenced EIP surveillance database
* Age greater than 2 days and younger than two months of age
* Resided in the catchment area on date of onset of their cough
* Born in a hospital in their state of residence
* ≥ 37 weeks of gestation at birth
* Not adopted, in foster care or living in a residential care facility
* Completed maternal interview
* Completed infant and maternal information

Controls were included if they met the following inclusion criteria:

* Age greater than 2 days and younger than 2 months of age on date of cough onset for the corresponding case infant
* Resided in the catchment area on date of cough onset for the corresponding case infant
* Born in a hospital in their state of residence
* ≥ 37 weeks of gestation at birth
* Not adopted, in foster care or living in a residential care facility
* Maternal interview completed
* Infant and maternal information complete

Exclusion Criteria:

Cases were excluded if they met any of the following exclusion criteria:

* Vaccination status of the mother unknown
* Infants whose mothers were vaccinated with Boostrix or an unknown vaccine brand

Controls were excluded if they met any of the following exclusion criteria:

* Vaccination status of the mother unknown
* A pertussis diagnosis prior to the cough onset date of the corresponding case infant
* Controls that were matched to Boostrix or an unknown brand cases

Ages: 2 Days to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants between 2 days to < 2 months of age for whom a case of pertussis was reported to one of 6 Emerging Infection Program (EIP) network sites included in the original Skoff et al. study (in 2017) and their respective control infants, for the study period.
Sampling Method: Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Number of pertussis cases in infants less than 2 months and matched controls | During the data collection period (from 01 January 2011 to 31 December 2014)
  Vaccine effectiveness at preventing pertussis in infants less than 2 months of age was estimated using conditional logistic regression.

SECONDARY OUTCOMES:
Number of pertussis cases requiring hospitalization in infants less than 2 months and matched controls | During the data collection period (from 01 January 2011 to 31 December 2014)
  Vaccine effectiveness at preventing pertussis requiring hospitalization was estimated using conditional logistic regression

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi Pasteur, Lyon, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Skoff TH, Blain AE, Watt J, Scherzinger K, McMahon M, Zansky SM, Kudish K, Cieslak PR, Lewis M, Shang N, Martin SW. Impact of the US Maternal Tetanus, Diphtheria, and Acellular Pertussis Vaccination Program on Preventing Pertussis in Infants <2 Months of Age: A Case-Control Evaluation. Clin Infect Dis. 2017 Nov 29;65(12):1977-1983. doi: 10.1093/cid/cix724. PMID 29028938
- [Result] Vargas-Zambrano JC, Clark LR, Johnson DR, Monfredo C, Pool V, Li L, Bouvet PE, Blangero Y, Macina D. Prenatal tetanus-diphtheria-acellular pertussis vaccine effectiveness at preventing infant pertussis. Vaccine. 2023 May 2;41(18):2968-2975. doi: 10.1016/j.vaccine.2023.03.048. Epub 2023 Apr 7. PMID 37032227